CLINICAL TRIAL: NCT02520960
Title: Pulmonary Vein Isolation for the Treatment of Paroxysmal Atrial Fibrillation by Combining the Analysis of the Unipolar Atrial Electrogram Modification With the Contact Force Sensing Technology: The Uniforce Study
Brief Title: Unipolar Atrial Electrogram Modification Combined to the Contact Force Sensing Technology for Pulmonary Vein Isolation
Acronym: Uniforce
Status: Completed | Type: Observational
Sponsor: Hôpital Privé Les Franciscaines (Other)
Collaborators: Clinique St Pierre, Perpignan, France (Unknown); Clinique Ambroise Paré, Neuilly sur Seine, France (Unknown); Hôpital Privé Clairval, Marseille, France (Unknown); Infirmerie Protestante de Lyon, Lyon, France (Ambiguous); Centre Hospitalo-Universitaire de Brabois, Vandoeuvre Les Nancy, France (Unknown); Centre Hospitalier Régional Universitaire Montpellier (Other); Paris Cardiovascular Research Center (Inserm U970) (Other Government); Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Agustin Bortone, MD, MD, Head of the Clinical Electrophysiology Unit, Hôpital Privé Les Franciscaines
Other Study IDs: 2014-30605
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: Catheter Ablation; Pulmonary Vein Isolation; Radiofrequency
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prospective observational multicentric study evaluating the efficacy of considering unipolar signal modification during radio frequency catheter ablation of patients with symptomatic paroxysmal atrial fibrillation in France between November 2013 and January 2015. All procedures were conducted according to the standard clinical care and current guidelines. Pulmonary vein isolation was guided according to force (at least 10 grams) and application vector (perpendicular to the wall) developed until the atrial unipolar electrogram recording became a complete positive signal. Patients were discharged from hospital free of any anti-arrhythmic drugs. Recurrence of arrhythmias at 12 months (primary outcome) was assessed by continuous 48-hour Holter at 1, 3, 6, 9 and 12 months post-catheter ablation.

DETAILED DESCRIPTION:
Patients and Setting: Consecutive patients referred to the participating institutions, from November 2013 to January 2015, for catheter ablation of symptomatic and drug resistant paroxysmal atrial fibrillation (AF) were enrolled in this observational 12-follow up study. Paroxysmal AF was defined as any episode of AF that terminates spontaneously in less than seven days. Eligibility criteria, as well as outcome measures have been detailed in other sections.

Radiofrequency catheter ablation for AF: All procedures were conducted according to the standard clinical care and North American and European guidelines. Of note, the investigators did not assign specific interventions to the subjects of the study, and all interventions (trans-oesophageal echocardiography, pulmonary vein isolation) are recommended by American Heart Association and European Society of Cardiology. AF catheter ablation were conducted under efficient vitamin K antagonists (INR 2-3) and general anesthesia without discontinuation of anti-arrhythmic drugs (AAD). Trans-esophageal echocardiography was performed for each patient within 48 hours before the procedure to exclude any intra-cardiac thrombi. Two long sheaths (Preface™, Biosense Webster, Diamond Bar, CA or SLO™, Saint Jude Medical, Minnetonka, MN) were advanced into the LA after two trans-septal punctures. Intravenous heparin was administered with a target activated clotting time beyond 320 seconds. Three catheters, inserted through the right femoral vein, were used for mapping and ablation: a 6F non deflectable hexapolar 2.5-2.5-2.5-2.5-247.5 mm interspacing electrodes catheter placed at the high right atrium (RA) or into the coronary sinus (CS) whenever possible (Curve: A-Josephson type, Biosense Webster), with its proximal electrode placed at the level of the inferior vena cava, a 7F circular decapolar mapping catheter (Lasso™) placed into the LA through one of the constantly perfused long sheaths and used to monitor PVI, and a 3.5 mm 7F externally irrigated-tip ablation contact force sensing catheter (SmartTouch™), placed within the LA through the second constantly irrigated long sheath. A LA anatomy shell was created with the aid of the Carto3 system (Biosense Webster). This shell was merged or not with 3D computed tomography scan acquired prior to the ablation procedure depending on operator's choice. Pulmonary veins were isolated two-by-two at their antral level by creating a continuous circular lesion. The carina regions were targeted only if PVs could not be isolated despite complete circular lesion creation around PVs ostia. Radiofrequency ablation settings used were: 30 W/48°C/17 ml per minute except for the posterior LA wall (25W/48°C/17 ml per min) and the ridge (35W/48°C/30 ml per min). Thirty minutes after PVI, entrance and exit blocks were rechecked for each PV. In case of PV reconnection, supplemental RF applications were performed in order to re-isolate PVs following a two-step approach.

Evaluation of the unipolar signal modification: every radiofrequency (RF) delivery was performed with a minimal 10 g of force, through the entire RF application and lasted 10 seconds after the unipolar atrial electrogram, recorded by the ablation catheter, which always demonstrated positive-negative morphology before ablation, became complete positive signal (except on the posterior LA wall where 5 supplemental seconds only were added). During individual RF applications, the modification of the unipolar atrial electrogram was monitored in real-time with the Carto™ system at a sweep speed of 200mm/s. Reference annotation signal was recorded from the bipolar signal of either electrodes 1-2 or 3-4 of the non-deflectable 6F hexapolar catheter, depending on whether the latter was placed into the CS or at the high RA. Unipolar signal was recorded from the 3.5mm distal electrode of the ablation catheter and was filtered on the Carto™ system with a [0.5-120] Hz band-pass filter and displayed in the Carto™ annotation viewer. The indifferent electrode was used as the cathode and was located at the level of the inferior vena cava.

Post-ablation Management and Follow-up: All patients were discharged home within 3 days, and enrolled in a 12-month follow-up. Post-procedure, AAD were discontinued while vitamin K antagonists were prescribed for 3 months. Subsequently, vitamin K antagonists were continued or not, depending on the CHA2DS2-VASc score of each patient. Patients were evaluated pre-discharge, at 1, 3, 6, 9 and 12 months post-procedure. Information collected included details of cardiac medications, NYHA functional class and history of any arrhythmias or other adverse events. In addition, a 12-lead ECG and 24-hour Holter monitoring were systematically obtained at each visit. Echocardiography was performed in all cases the day after procedure. No antiarrhythmic medication was prescribed following ablation. If there was documented recurrence of symptomatic AF during the 3-month blanking period and the patient required antiarrhythmic drug therapy, a previously ineffective but tolerated class 1 or class 3 (sotalol) drug was the preferred option. Atrial tachycardia/AF recurrence was considered, any episode lasting > 30 s (either symptomatic or asymptomatic) subsequent to a 3-month blanking period.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal symptomatic and drug resistant atrial fibrillation (AF). Paroxysmal AF was considered any episode of AF that terminates spontaneously in less than seven days.

Exclusion Criteria:

* age <18 or >80 year-old
* left atrial volume >200 ml
* presence of a mechanical mitral valve prosthesis
* impaired thyroid function
* left ventricular ejection fraction <40%
* patient under guardianship
* contraindication to anticoagulant therapy
* current malignancy
* prior catheter or surgical AF ablation
* persistent or long-standing persistent AF

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients referred to the participating institutions, from November 2013 to January 2015, for catheter ablation of symptomatic and drug resistant PAF. Paroxysmal AF was considered any episode of AF that terminates spontaneously in less than seven days.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Recurrence of Atrial Arrhythmias | 12 months

SECONDARY OUTCOMES:
Frequency of Pulmonary Vein Reconnection | 30 mins
  Recurrence of the electrical conduction between atria and pulmonary veins

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Bortone, MD, Principal Investigator — Service de Cardiologie, Hôpital Privé Les Franciscaines, Nîmes, France
Locations (1):
- Hôpital Privé Les Franciscaines, Nîmes, France

REFERENCES:
- [Result] Bortone A, Brault-Noble G, Appetiti A, Marijon E. Elimination of the negative component of the unipolar atrial electrogram as an in vivo marker of transmural lesion creation: acute study in canines. Circ Arrhythm Electrophysiol. 2015 Aug;8(4):905-11. doi: 10.1161/CIRCEP.115.002894. Epub 2015 Jun 19. PMID 26092576
- [Result] Bortone A, Appetiti A, Bouzeman A, Maupas E, Ciobotaru V, Boulenc JM, Pujadas-Berthault P, Rioux P. Unipolar signal modification as a guide for lesion creation during radiofrequency application in the left atrium: prospective study in humans in the setting of paroxysmal atrial fibrillation catheter ablation. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1095-102. doi: 10.1161/CIRCEP.113.000749. Epub 2013 Oct 4. PMID 24097371
- [Derived] Bortone A, Lagrange P, Cauchemez B, Durand C, Dieuzaide P, Prevot S, Mechulan A, Pambrun T, Martin R, Parlier P, Masse A, Marijon E, Albenque JP. Elimination of the negative component of the unipolar electrogram as a local procedural endpoint during paroxysmal atrial fibrillation catheter ablation using contact-force sensing: the UNIFORCE study. J Interv Card Electrophysiol. 2017 Sep;49(3):299-306. doi: 10.1007/s10840-017-0264-4. Epub 2017 Jun 22. PMID 28643171